CLINICAL TRIAL: NCT02416401
Title: Attention Training for Learning Enhancement and Resilience Trial
Acronym: ALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Iowa (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1006-14
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Age-related Cognitive Decline
Keywords: healthy; aging; cognition; age-related cognitive decline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 36 treatment sessions, 4-5 times weekly, one hour each session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 36 treatment sessions, 4-5 times weekly, one hour each session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Arms: Experimental Treatment
Other: Commercially available computerized training
  Arms: Active Comparator

SUMMARY:
Healthy aging is associated with a decline in multiple cognitive domains, as well as motor control function. The long-term consequences of cognitive and functional impairment resulting from age-related cognitive decline are well documented in the scientific and clinical literature, with significant evidence of related problems with independent functional abilities. This study aims to understand how the experimental computer program can affect cognition and attention in participants with age-related cognitive decline.

DETAILED DESCRIPTION:
Following consent, participants will engage in an assessment process to determine eligibility. Once eligibility is confirmed, participants will be scheduled for another assessment session to determine current level of cognitive function. This process consists of paper-pencil surveys and computerized tests. Following the assessment process, participants will engage in an Internet browser-delivered training sessions conducted on any internet-accessible computer. The computerized training sessions can be done up to 7 times a week (once a day) or at the participant's convenience (the recommended time commitment is 5 times a week). Following the completion of training, the participant's cognitive function will be re-assessed. Participation is voluntary and participants may withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 65 years of age or older
* Participants must have a diagnosis of age-related cognitive decline as confirmed by interview and performance on screening assessments
* Participants must be fluent English speakers
* Participants must have adequate visual, auditory, and motor capacity to use computerized intervention

Exclusion Criteria:

* Participants with diagnosis of PTSD, depression or other psychologically diagnosable emotional disorder
* Participants with a history of conditions that could affect thinking abilities, including brain injury, mental illness, cancer, or other neurological conditions (multiple sclerosis, seizure disorder), HIV/AIDS will be excluded
* Participants enrolled in another concurrent research study will be excluded
* Participants who have difficulty performing assessments or comprehending or following spoken instructions, in the judgment of the screening clinician, will be excluded
* Participants with a current or significant past history of substance abuse will be excluded
* Participants who show signs of suicidal ideations or behaviors will be excluded and referred for appropriate treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Attention Measures aimed to test attention | 6 months
  Measures aimed to test attention
Executive Function | 6 months
  Tasks targeting inhibitory control
Functional Capacity | 6 month
  Performance on directly observable functional measure

SECONDARY OUTCOMES:
Quality of Sleep | 6 months
  assessing sleep quality

OTHER OUTCOMES:
Quality of life | 6 months
  Assessments and questionnaire assessing quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Harvard Medical School, Boston, Massachusetts

REFERENCES:
- [Background] Gazzaley A, Cooney JW, Rissman J, D'Esposito M. Top-down suppression deficit underlies working memory impairment in normal aging. Nat Neurosci. 2005 Oct;8(10):1298-300. doi: 10.1038/nn1543. Epub 2005 Sep 11. PMID 16158065
- [Background] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038
- [Background] Burke SN, Barnes CA. Neural plasticity in the ageing brain. Nat Rev Neurosci. 2006 Jan;7(1):30-40. doi: 10.1038/nrn1809. PMID 16371948
- [Background] Cicerone KD, Dahlberg C, Malec JF, Langenbahn DM, Felicetti T, Kneipp S, Ellmo W, Kalmar K, Giacino JT, Harley JP, Laatsch L, Morse PA, Catanese J. Evidence-based cognitive rehabilitation: updated review of the literature from 1998 through 2002. Arch Phys Med Rehabil. 2005 Aug;86(8):1681-92. doi: 10.1016/j.apmr.2005.03.024. PMID 16084827
- [Derived] VanVleet T, Voss M, Dabit S, Mitko A, DeGutis J. Randomized control trial of computer-based training targeting alertness in older adults: the ALERT trial protocol. BMC Psychol. 2018 May 3;6(1):22. doi: 10.1186/s40359-018-0233-4. PMID 29724228